CLINICAL TRIAL: NCT00355589
Title: A Randomized, Double-Blind, Multicenter, Parallel Study Evaluating the Efficacy and Safety of a Combination of Ramipril Plus Hydrochlorothiazide Versus the Component Monotherapies in Subjects With Essential Hypertension
Brief Title: Ramipril and Hydrochlorothiazide Alone and in Combination for the Treatment of Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K749-06-3001; B5051001 (Other: Pfizer)
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension; Blood Pressure, High
Keywords: Hypertension; High Blood Pressure; Diuretic; Angiotensin converting enzyme inhibitor; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Hydrochlorothiazide

INTERVENTIONS:
Drug: Ramipril and hydrochlorothiazide

SUMMARY:
The purpose of this study is to determine if there is greater blood pressure reduction using ramipril or hydrochlorothiazide alone or ramipril and hydrochlorothiazide together.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed, or newly diagnosed essential hypertension. Blood pressure must be within a minimum and maximum range prior to drug treatment.

Exclusion Criteria:

* Inability to discontinue all prior antihypertensive medications
* Heart failure
* History of stroke, myocardial infarction, or chest pain within 3 years, or an abnormal heart rhythm
* Liver or kidney disease
* Certain drugs used to treat other conditions like an enlarged prostate gland, or arthritis
* Allergy or reactions to certain medications used to treat high blood pressure

Other protocol-defined inclusion and exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Compare the effects on sitting diastolic blood pressure of two antihypertensive drugs in combination against each antihypertensive alone after an eight week treatment period.

SECONDARY OUTCOMES:
Compare the effect on sitting diastolic blood pressure of two antihypertensive drugs in combination taken once daily against one antihypertensive drug taken twice daily.
Compare the effect on sitting diastolic blood pressure of a dose of an antihypertensive drug taken once daily against half of the same dose taken twice daily.
Compare the effect on the sitting and standing blood pressure among all treatment groups.
Compare the safety of each medication regimen stated above.
Compare the effect on mean 24-hour diastolic blood pressure (ABPM) of the medication regimens stated above.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Cahaba Research Inc., Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Pulmonary Associates, Glendale, Arizona
  - Impact Clinical Trials, Beverly Hills, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Marin Endocrine Care and Research, Greenbrae, California
  - Memorial Research Medical Clinic, Long Beach, California
  - The Intermed Group; Samaritan Medical Tower, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Clinical Trials Research, Roseville, California
  - Bayview Research Group, Studio City, California
  - Viking Clinical Research, Temecula, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - University Clinical Research Deland, Inc., DeLand, Florida
  - South Florida Clinical Research Center, Hollywood, Florida
  - Innovative Research of West Florida, Largo, Florida
  - International Research Associates, LLC, Miami, Florida
  - Lifespan Research Foundation, Miami, Florida
  - Sun Coast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Executive Health and Research Associates, Inc., Atlanta, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - James R. Herron, MD, Ltd., Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Michigan Institute of Medicine, Livonia, Michigan
  - Medical Research Associates, Traverse City, Michigan
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Partners in Primary Care, Voorhees Township, New Jersey
  - Cumberland Research Assocites, LLC, Fayetteville, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - The Lipid Center, Statesville, North Carolina
  - Lyndhurst Gynecologic Associates, PA, Winston-Salem, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Sterling Research Group, Inc., Cincinnati, Ohio
  - Smith Clinical Research, Marion, Ohio
  - Radiant Research - Mogadore, Mogadore, Ohio
  - Lion Research, Norman, Oklahoma
  - Medford Medical Clinic Research Dept., Medford, Oregon
  - Philadelphia Health Associates, Philadelphia, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Radiant Research - Greer, Greer, South Carolina
  - MetaClin Research, Inc., Austin, Texas
  - Punzi Medical Center, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - WellMed Medical Management, San Antonio, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - The Chase Wellness Center, Inc, Virginia Beach, Virginia
  - Radiant Research - Tacoma, Lakewood, Washington

REFERENCES:
- [Derived] White WB, Cleveland JM, Rolleri RL; Ramipril-Hydrochlorothiazide Study Group. Utility of semiautomatic clinic and 24-h ambulatory blood pressure measurements to evaluate combination therapy: the Ramipril-Hydrochlorothiazide Hypertension trial. J Hum Hypertens. 2008 Aug;22(8):559-68. doi: 10.1038/jhh.2008.26. Epub 2008 May 8. PMID 18463672